CLINICAL TRIAL: NCT02194595
Title: Preserving Beta-cell Function in Type 2 Diabetes With Exenatide and Insulin (PREVAIL)
Acronym: PREVAIL
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Mount Sinai Hospital, Canada (Other)
Collaborators: Canadian Institutes of Health Research (CIHR) (Other Government); University of Toronto (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 14-0128-A
Record Dates: First submitted 2014-07-16; First posted 2014-07-18 (Estimated); Last update posted 2022-04-11 (Actual); Status verified 2022-04

CONDITIONS: Type 2 Diabetes
Keywords: type 2 diabetes; beta-cell function; GLP-1; insulin
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Insulin Resistance | interventions — Exenatide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Basal insulin and exenatide (Experimental): Participants in this arm will undergo an 8-week course of treatment with exenatide and insulin glargine. Exenatide will be initiated at 5ug subcutaneous (sc) bid (before breakfast and before dinner) for the first 4 weeks, followed by 10ug bid for the next 4 weeks. Glargine sc injection at bedtime will be titrated to fasting glucose.
  Interventions: Drug: Basal insulin and exenatide
- Basal insulin only (Active Comparator): Participants in this arm will undergo an 8-week course of treatment with glargine sc injection at bedtime, titrated to target fasting glucose.
  Interventions: Drug: Basal insulin only
- Basal Insulin and bolus insulin (Active Comparator): Participants in this arm will undergo an 8-week course of multiple daily insulin injection therapy, consisting of titrated basal insulin glargine at bedtime and insulin lispro before each meal.
  Interventions: Drug: Basal insulin and bolus insulin

INTERVENTIONS:
Drug: Basal insulin and exenatide
  Other Names: Basal insulin glargine; Exenatide
  Arms: Basal insulin and exenatide
Drug: Basal insulin only
  Other Names: Basal insulin glargine
  Arms: Basal insulin only
Drug: Basal insulin and bolus insulin
  Other Names: Basal insulin glargine; Pre-meal insulin lispro
  Arms: Basal Insulin and bolus insulin

SUMMARY:
Type 2 diabetes mellitus is a chronic metabolic disorder characterized by progressive deterioration in the function of the pancreatic beta-cells, which are the cells that produce and secrete insulin (the hormone primarily responsible for the handling of glucose in the body). The investigators propose a randomized controlled trial to determine whether combining basal insulin with a new medication called exenatide is a therapeutic strategy that can preserve beta-cell function early in the course of type 2 diabetes.

DETAILED DESCRIPTION:
In this open-label, parallel-arm randomized controlled trial, adults with T2DM of ≤7 years duration on 0-2 anti-diabetic medications will be randomized to 8-weeks treatment with either (i) basal insulin glargine, (ii) intensive insulin therapy consisting of glargine and pre-meal insulin lispro, or (iii) glargine and the GLP-1 agonist exenatide (twice daily). They will then go into a 12-week washout on lifestyle modification only. Beta-cell function will be assessed by determining the Insulin Secretion-Sensitivity Index-2 (ISSI-2) on oral glucose tolerance test (OGTT) performed at baseline, 4-weeks, 8-weeks, and 20-weeks. The primary outcome will be mean beta-cell function (ISSI-2) over the 8-week treatment period.

ELIGIBILITY:
Inclusion Criteria:

1. Men and women between the ages of 30 and 80 years inclusive
2. T2DM diagnosed by a physician ≤7 years prior to enrolment
3. On 0-2 anti-diabetic medications, with no change in dose/regimen in the preceding 4 weeks
4. A1c at screening between 5.5% and 9.0% inclusive if on anti-diabetic medications, or between 6.0% and 9.5% inclusive if on no oral anti-diabetic medication
5. BMI ≥ 23 kg/m2
6. Negative pregnancy test at recruitment for all women with childbearing potential

Exclusion Criteria:

1. Current anti-diabetic treatment with insulin or a glucagon-like peptide-1 (GLP-1) agonist
2. Type 1 diabetes or secondary forms of diabetes
3. History of hypoglycemia unawareness or severe hypoglycemia requiring assistance
4. Hypersensitivity to insulin, exenatide, or the formulations of these products
5. Renal dysfunction as evidenced by estimated glomerular filtration rate (eGFR)<30 ml/min by Modification of Diet in Renal Disease (MDRD) formula
6. History of pancreatitis
7. Family or personal history of Multiple Endocrine Neoplasia type 2 (MEN-2) or familial medullary thyroid carcinoma (MTC)
8. Personal history of non-familial medullary thyroid carcinoma (MTC)
9. Malignant neoplasm requiring chemotherapy, surgery, radiation or palliative therapy within the previous 5 years (with the exception of basal cell skin cancer)
10. Unwillingness to perform capillary glucose monitoring at least 4 times a day during treatment
11. Pregnancy or unwillingness to use reliable contraception. Women should not be planning pregnancy for the duration of the study or the first 3 months after the study. Reliable contraception includes birth control pill, intra-uterine device, abstinence, tubal ligation, partner vasectomy, or condoms with spermicide.
12. Any factor likely to limit adherence to the protocol, in the opinion of investigator

Ages: 30 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 105 (Actual)
Dates: Start 2014-09; Primary Completion 2021-12 (Actual); Study Completion 2022-02 (Actual)

PRIMARY OUTCOMES:
Mean beta-cell function over the 8-week treatment period, measured using the Insulin Secretion-Sensitivity Index-2 (ISSI-2) | 8 weeks
  ISSI-2 is an established measure of beta-cell function. ISSI-2 is defined as the product of (i) insulin secretion measured by the ratio of the area-under-the-insulin-curve to the area-under-the-glucose curve and (ii) insulin sensitivity measured by the Matsuda index. The primary outcome comparison is between the glargine/exenatide and glargine only arms.

SECONDARY OUTCOMES:
Baseline-adjusted beta-cell function at 20 weeks | 20 weeks
  The secondary outcome of baseline-adjusted beta-cell function at 20 weeks will be measured with the Insulin Secretion-Sensitivity Index-2 (ISSI-2)
Baseline-adjusted glycemic control at 20 weeks | 20 weeks
  The secondary outcome of baseline-adjusted glycemic control at 20 weeks will be assessed by A1c (glycated hemoglobin)
Endothelial function at 8 weeks | 8 weeks
  Endothelial function will be assessed as the digital endothelial vasomotor function in response to reactive hyperemia using pulse amplitude tonometry, which will be measured by the pulse amplitude response to hyperemia (PAT ratio)
Baseline-adjusted glycemic control at 8 weeks | 8 weeks
  Baseline-adjusted glycemic control at 8 weeks will be measured by A1c

OTHER OUTCOMES:
Baseline-adjusted insulin sensitivity at 8 weeks | 8 weeks
  Baseline-adjusted insulin sensitivity at 8 weeks will be measured by Matsuda index
Baseline-adjusted insulin sensitivity at 20 weeks | 20 weeks
  Baseline-adjusted insulin sensitivity at 20 weeks will be measured by Matsuda index

CONTACTS AND LOCATIONS:
Overall Officials: Ravi Retnakaran, MD, Principal Investigator — MOUNT SINAI HOSPITAL
Locations (1):
- Mount Sinai Hospital, Toronto, Ontario, Canada

REFERENCES:
- [Derived] Retnakaran R, Pu J, Ye C, Emery A, Kramer CK, Zinman B. The vascular function effects of adding exenatide or meal insulin to basal insulin therapy in early type 2 diabetes. Cardiovasc Diabetol. 2023 Mar 9;22(1):50. doi: 10.1186/s12933-023-01781-z. PMID 36894921